CLINICAL TRIAL: NCT03609060
Title: A Phase II Study of Dexamethasone Added to Induction and Post-remission Therapy in Older Patients with Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Dexamethasone Added to Intensive Chemotherapy in Older Patients with Acute Myeloid Leukemia (AML)
Acronym: DEXAML-02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEXAML-02 (LAM-SA 2018)
Record Dates: First submitted 2018-06-28; First posted 2018-08-01 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Elderly patients
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEXAML (Experimental): Induction therapy:
  Idarubicin 8 mg/m²/day, IV over 15 minutes, D1 to D5 + Cytarabine 100 mg/m²/d, IV continuous 24h-infusion D1 to D7 + Lomustine 200 mg/m²/d, orally at D1 + Dexamethasone 10 mg/12h, IV over 30 minutes, D1 to D3. Addition of midostaurin in patients with Fms-like tyrosine kinase 3-internal tandem ( FLT3-ITD) or Fms-like tyrosine kinase 3-tyrosine kinase domain (FLT3-TKD) mutations is allowed.
  Post remission therapy:
  Idarubicin 8 mg/m², IV over 15 minutes, D1 + Cytarabine 50 mg/m²/12h, subcutaneous, D1 to D5 + Dexamethasone 20 mg/d, IV over 30 minutes, D1. Addition of midostaurin in patients with FLT3-ITD or FLT3-TKD mutations is allowed. Intermediate dose cytarabine is allowed for patients with Core Binding Factor AML (CBF-AML).
  Allogeneic stem-cell transplantation allowed after 2 to 4 cycles
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10 mg/12h, IV over 30 minutes, D1 to D3 concomitant to induction and post remission chemotherapy in elderly patients with AML Induction

SUMMARY:
Recent preclinical and clinical data strongly suggested that dexamethasone could improve the activity of intensive chemotherapy in AML. In this study, the FILO study group will assess the impact of adding dexamethasone to both induction and consolidation therapy in older AML patients with intermediate or favorable risk.

DETAILED DESCRIPTION:
Patients will receive dexamethasone in addition to induction and post-remission chemotherapy

The principal objective of the study is to determine whether adding dexamethasone to induction and post-remission therapy results in significant improvement of event-free survival (EFS) as compared with an historical cohort of the FILO LAM-SA 2007 trial.

Induction therapy: Idarabucin + Cyrarabine + Lomustine (ICL) + Dexamethasone. Idarubicin 8 mg/m²/day, IV over 15 minutes, D1 to D5; Cytarabine 100 mg/m²/d, IV continuous 24h-infusion D1 to D7; Lomustine 200 mg/m²/d, orally at D1; Dexamethasone 10 mg/12h, IV over 30 minutes, D1 to D3.

Post remission therapy: Idarabucin + Cyrarabine (IC) + Dexamethasone

Idarubicin 8 mg/m², IV over 15 minutes, D1; Cytarabine 50 mg/m²/12h, subcutaneous, D1 to D5; Dexamethasone 20 mg/d, IV over 30 minutes, D1.

ELIGIBILITY:
Inclusion Criteria:

1. > 60 years of age.
2. Newly diagnosed AML according to the World Health Organization (WHO) 2016 either de novo AML or therapy-related AML (i.e AML arising after previous cytotoxic therapy or radiation)
3. AML with favorable or intermediate cytogenetic risk according to Medical Research Council (MRC 2010) classification.
4. Subjects should be eligible for intensive chemotherapy by Idarubicin, cytarabine, Lomustine.
5. Eastern Cooperative Oncology Group (ECOG) performance status < 3 (appendix 1).
6. SORROR score ≤ 3 (appendix 2).
7. Adequate baseline organ function defined by the criteria below:

   * Total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) unless bilirubin rise is due to Gilbert's syndrome
   * Alanine Aminotransferase (ALAT) and Aspartate Transaminase (ASAT) ≤ 3xULN
   * creatinin clearance (Cockcroft-Gault) ≥ 30 ml/min
   * Unless considered due to leukemic organ involvement
8. Adequate cardiac function with Left Ventricular Ejection Fraction (LVEF) ≥50%
9. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
10. Women will be menopausal to be enrolled
11. The patient must give written (personally signed and dated) informed consent before completing any study-related procedure which means assessment or evaluation that would not form part of the normal medical care of the patient and before the start of induction chemotherapy.
12. Affiliated to the French Social Security (Health Insurance).

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL) or acute megakaryocytic leukemia (AML-FAB M7).
2. AML with adverse cytogenetic risk according to the MRC 2010 classification.
3. AML arising from myelodysplastic syndromes, myeloproliferative disorders or chronic myelo-monocytic leukemia according to WHO classification (2016).
4. AML with Philadelphia chromosome or with BCR-ABL1.
5. Known active central nervous system leukemia
6. Previous anti-AML treatment other than hydroxyurea.
7. Cumulative anthracycline dose equivalent to ≥550 mg/m².
8. Treatment with an investigational drug within 30 days or 5 half-life whichever is longer, preceding the first dose of study medication.
9. Prior history of cancer unless controlled for at least 2 years and except for basal cell carcinoma, non-melanoma skin cancer and in situ cervical carcinoma.
10. Severe medical or mental condition precluding the administration of protocol treatments
11. Any sign of active uncontrolled disease including but not restricted to cardiac disease, infections, hepatitis.
12. Any severe chronic disease potentially interfering with the protocol including HIV infection, active hepatitis B or C.
13. Any severe conditions inducing contra-indications to dexamethasone including uncontrolled diabetes, infections, hypertension, stomach ulcer, mental illness, myasthenia or glaucoma.
14. Any serious medical condition, laboratory abnormality, or psychiatric illness that would place the participant at an unacceptable risk or prevent them from giving informed consent.
15. Known active HIV, Hepatitis B or C infection.
16. Pregnancy or breastfeeding.
17. Patients who are incapacitated, under wardship, legal guardianship, or under the protection of the courts.
18. Patients under State Medical Assistance (AME).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Event Free survival (EFS) | Within 2 years after the start of the Treatement
  Time from the date of induction start to the date of induction failure, relapse from CR or CRi, or death from any cause, whichever occurs first. CR, CRi, relapse from CR or CRi and induction failure are defined according to the ELN 2017 recommendations

SECONDARY OUTCOMES:
Treatment response | Up to 45 day
  Response to therapy after induction therapy defined as CR or CRi according to the 2017 European Leukemia Net (ELN) recommendations.
Minimal Residual Disease (MRD) | Up to day 45 after induction chemotherapy, second and last consolidation cycle.
  Presence of MRD after induction therapy and after post-remission therapy, measured by either quantitative PCR or flow cytometry
Allogenic Stem Cells Transplantation (ASCT) | Up to one year
  Number of patients with ASCT
Remission duration (relapse from CR or CRi) | two years
  Time from the date of CR or CRi to the date of relapse according to the 2017 ELN recommendations
Relapse Free Survival (RFS) | two years
  Time from the date of CR or CRi to the date of relapse or death from any cause, whichever occurs first, according to the ELN 2017 recommendations
Overall Survival (OS) | two years
  Time from the date of randomization to the date of death from any cause
Adverse events | up to 60 months
  Incidence and severity of Adverse Events according to the descriptions and grading scale found in the National Cancer Institute - Common Terminology Criteria (NCI-CTC) criteria v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Christian RECHER, MD PD, Principal Investigator — +33 5 31 15 63 55
Locations (25):
- France (25):
  - CHU ANGERS - Maladies du sang, Angers
  - Ch Avignon, Avignon
  - CH de la Côte Basque - Hématologie, Bayonne
  - CHRU JEAN MINJOZ - Hématologie, Besançon
  - CH de Béziers - Hématologie, Béziers
  - CHU Brest - Hôpital Morvan - Hématologie Clinique, Brest
  - Clinique du Parc - Hématologie, Castelnau-le-Lez
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - CHU Grenoble - Hématologie Clinique, Grenoble
  - Institut Paoli-Calmettes - Hématologie 2, Marseille
  - CHR de Mercy - Hématologie, Metz
  - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - HOPITAL E. MULLER - Hématologie, Mulhouse
  - CHU HOTEL DIEU - Hématologie Clinique, Nantes
  - CHR ORLEANS - Hématologie, Orléans
  - HOPITAL COCHIN - Hématologie, Paris
  - CENTRE HOSPITALIER SAINTJEAN - Hématologie Clinique, Perpignan
  - Hôpital Haut Levêque- CFM -Hématologie Clinique Et Thérapie Cellulaire, Pessac
  - CHU La Milétrie - Hématologie Clinique, Poitiers
  - CHU Reims - Hôpital Robert Debré - Hématologie Clinique, Reims
  - CHU Pontchaillou - Hématologie, Rennes
  - CHU Hautepierre - Hématologie, Strasbourg
  - Institut Universitaire du Cancer de Toulouse Oncopole - Service d'Hématologie, Toulouse
  - CHU Bretonneau - Centre Henri Kaplan - Hématologie et Thérapie Cellulaire, Tours
  - CHU Nancy - Hopitaux Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- See also: FILO Internet site — http://www.filo-leucemie.org